CLINICAL TRIAL: NCT00513383
Title: Phase I Study Panitumumab Plus Chemoradiotherapy and Induction Chemotherapy in Patients With Locally Advanced Squamous Cell Cancer of the Head and Neck
Brief Title: Panitumumab Chemoradiotherapy Chemotherapy for Squamous Cancer of the Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Amgen (Industry)
Responsible Party: Principal Investigator, Lori J. Wirth, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-401
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: basaloid squamous cell carcinoma; undifferentiated carcinoma; adenosquamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma; Carcinoma, Adenosquamous | interventions — Panitumumab; Carboplatin; Paclitaxel; Radiotherapy, Intensity-Modulated; Fluorouracil; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A (Experimental): Determine the best dosing of panitumumab, chemotherapy and radiation.
  Interventions: Drug: Panitumumab; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Intensity Modulated Radiation Therapy
- Part B (Experimental): Determine the best dosing of induction chemotherapy combined with panitumumab prior to receiving panitumumab and chemoradiotherapy.
  Interventions: Drug: Panitumumab; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Intensity Modulated Radiation Therapy; Drug: 5-Fluorouracil; Drug: Docetaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Panitumumab — Part A: Intravenously once a week for 7 weeks Part B (Induction Chemotherapy): Intravenously on Day 1 of a 21-day cycle for 3 cycles Part B (After Induction chemotherapy): Intravenously once a week for 7 weeks at the dosing level established during Part A
Drug: Carboplatin — Part A: Intravenously once weekly for 7 weeks Part B (Following induction therapy): Intravenously once a week for 7 weeks
Drug: Paclitaxel — Part A: Intravenously once weekly for 7 weeks Part B (Following induction therapy): Intravenously once a week for 7 weeks
Radiation: Intensity Modulated Radiation Therapy — Part A: Daily five days a week for 7 weeks Part B (After Induction therapy): Daily five days a week for 7 weeks
  Other Names: IMRT
Drug: 5-Fluorouracil — Intravenously at one of two dose levels on days 1-4 of a 21-day cycle for three cycles
  Other Names: 5-FU
  Arms: Part B
Drug: Docetaxel — Intravenously on day 1 of a 21-day cycle for 3 cycles
  Arms: Part B
Drug: Cisplatin — Intravenously on day 1 of a 21-day cycle for 3 cycles
  Arms: Part B

SUMMARY:
This study is being done to test whether panitumumab, in combination with chemotherapy and radiation is safe in people with head and neck cancer. Another goal of this study is to find the highest dose of the study drugs that can be given safely without causing serious sife effects. Panitumumab is a type of drug called a monoclonal antibody that has been studied in other types of cancers, such as kidney and colon. This monoclonal antibody is directed against the epidermal growth factor receptor (EGFR). EGFR has been found on the majority of head and neck cancer cells. By blocking EGFR, this monoclonal antibody may inhibit the growth of head and neck cancer cells.

DETAILED DESCRIPTION:
* There are two parts to this study: Part A and Part B. Participants enrolled in Part A of this study received panitumumab and chemoradiotherapy. Participants enrolled in Part B will receive panitumumab in combination with induction chemotherapy followed by chemoradiotherapy.
* The main purpose of Part A was to examine the safety and the best dosing of panitumumab, chemotherapy and radiation for the treatment of head and neck cancer. The best dosing was determined by increasing doses of chemotherapy given in combination with panitumumab during radiation. The chemotherapy drugs being used in Part A were carboplatin and paclitaxel, which are standard therapies used in head and neck cancer. These drugs were be added to radiation and this combination is called chemoradiotherapy. The investigators have determined the best dose of panitumumab and chemotherapy to give with radiation, Part B has now begun.
* The main purpose of Part B is to examine the safety and best dosing of chemotherapy combined with panitumumab (called induction therapy) prior to receiving panitumumab and chemoradiotherapy. The drugs that are used for induction chemotherapy will be docetaxel, cisplatin and 5-fluorouracil. These drugs are also standard therapies used in head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven squamous cell carcinoma of the head and neck or its variants (such as basaloid squamous cell carcinoma, undifferentiated carcinoma, or adenosquamous cell carcinoma). Primary tumor sites eligible include: nasopharynx, oral cavity, oropharynx, hypopharynx, larynx or unknown primary SCCHN
* Stage III or IV disease, without evidence of distant metastasis, according to American Joint Committee on Cancer
* Measurable disease, according to RECIST.
* No prior chemotherapy, radiotherapy or attempted complete resection of the SCCHN. Diagnostic biopsy, including excisional nodal biopsy and/or tonsillectomy is allowed if the subject has measurable disease at the time of enrollment
* 18 years of age or older
* ECOG Performance Status of 0 or 1
* No active alcohol addiction or other condition that, in the opinion of the study investigators, would interfere with the subject's ability to comply with the treatment plan
* Adequate hepatic and renal function
* Women of childbearing potential must have a negative pregnancy test within 2 weeks of study entry.

Exclusion Criteria:

* Pregnant or breast feeding women
* Symptomatic peripheral neuropathy of grade 2 or higher by NCI CTCAEv3.0
* Grade 3 or more hearing loss
* History of other malignancy within the previous 5 years, except for nonmelanoma skin cancer, carcinoma in situ of the cervix, bladder or head and neck
* Prior radiation to head and neck
* Other serious illness or medical conditions
* Patients who experienced an involuntary weight loss of more than 20% of their body weight in the 2 months preceding study entry
* Concurrent treatment with any other anticancer therapy
* Prior therapy which affects or targets the ErbB pathway, including any inhibitors of EGFR and ErbB2
* Participation in an investigational drug trial within 30 days of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-04; Primary Completion 2010-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To identify the maximally tolerated dose of paclitaxel given with panitumumab plus carboplatin chemoradiotherapy. | 2 years
To identify the maximally tolerated dose or biologically acceptable dose of TPF, varying the 5-FU dose, given with a fixed dose of panitumumab, prior to concurrent carboplatin, paclitaxel, panitumumab chemoradiotherapy. | 2 years

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of the combination of Pan-CRT and Pan-TPF. | 2 years
To estimate the overall response rate to Pan-TPF. | 2 years
To estimate the overall response rate of sequential therapy. | 2 years
To estimate the rate of pathologic complete response of primary tumor biopsy, to estimate 2-year disease free survival and overall survival.
To evaluate functional outcome at 2 years with respect to speech, swallowing and overall quality of life. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lori J. Wirth, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Wirth, L.J. Phase I Study of Panitumumab, Chemotherapy, and Intensity-modulated Radiotherapy (IMRT) for head and neck cancer (HNC). Abstract-No.6083 2007 ASCO Annual Meeting